CLINICAL TRIAL: NCT03380000
Title: Acute Blood Pressure-lowering Effects of Beetroot Juice in Postmenopausal Women With and Without Hypertension
Brief Title: Effect of Beetroot Juice on Blood Pressure Regulation in Post Menopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, David N. Proctor, PhD, Professor of Kinesiology, Physiology, and Medicine, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 00043633
Record Dates: First submitted 2017-12-10; First posted 2017-12-20 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Postmenopausal Women
Keywords: Dietary nitrate supplementation; Beetroot juice

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Treatment order will be randomly assigned to participants by Clinical Research Center (CRC) staff using computer-based mathematical software. The generated list that determines each participants treatment order will be kept in a secure location in the CRC which cannot be accessed directly by research team members.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitrate rich beetroot juice (Active Comparator): Subjects will consume 140 ml of beetroot juice (Beet-It Organic Shot) approximately 90 min before physiological testing.
  Interventions: Drug: Beetroot juice
- Nitrate depleted beetroot juice (Placebo Comparator): Subjects will consume 140 ml of beetroot juice (Beet-It Organic Placebo) approximately 90 min before physiological testing.
  Interventions: Drug: Beetroot juice placebo

INTERVENTIONS:
Drug: Beetroot juice — This beverage contains 0.3 g of inorganic nitrate per 70 ml container, and is bottled and supplied by James White Drinks (UK).
  Other Names: Beet-It Organic Shot
  Arms: Nitrate rich beetroot juice
Drug: Beetroot juice placebo — This beverage is identical in look and taste to the Beet-It organic shot, but has the nitrate removed. It is also bottled and supplied by James White Drinks (UK).
  Other Names: Beet-It Organic placebo
  Arms: Nitrate depleted beetroot juice

SUMMARY:
In this study the investigators will test the hypothesis that acute consumption of inorganic nitrate (supplied in concentrated beetroot juice) reduces artery stiffness and resting blood pressure, and lessens the rise in blood pressure during handgrip exercise in postmenopausal women. Understanding and improving artery function and blood pressure regulation in women is important because they undergo accelerated arterial stiffening after menopause and have much larger increases in blood pressure when they exercise compared with either premenopausal women or men of similar age.

DETAILED DESCRIPTION:
Postmenopausal women have stiff central arteries and exaggerated blood pressure (BP) responses during exercise compared with either premenopausal women or men of similar age. Arterial stiffness and exaggerated BP responses to exercise are prognostic for heart wall thickening, future hypertension, adverse cardiovascular events, and mortality. Previous studies have reported that acute consumption of nitrate-rich beetroot juice can lower resting and exercising BP responses in older adults. However, these studies included both sexes and did not compare the effects of beetroot juice to a nitrate-depleted placebo (a true control). Thus, the potential BP lowering effects of nitrate supplementation per se have not been established in postmenopausal women. The present study examines the acute (single dose) effects of nitrate-rich beetroot juice on resting hemodynamics (peripheral and central BP, arterial wave properties, etc), and physiological responses to handgrip exercise in metabolically healthy post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Resting systolic blood pressure less than or equal to 160 mmHg
* Resting diastolic blood pressure less than or equal to 100 mmHg

Exclusion Criteria:

* Overt cardiovascular, metabolic, hematologic, pulmonary, renal, musculoskeletal, and/or neurological disease(s)
* Users of any tobacco and/or nicotine products (smokers, chewing tobacco, nicotine-containing patches/gum, smokeless cigarettes)
* Body mass index greater than 35
* Total cholesterol greater than 239 mg/dl
* LDL cholesterol greater than 159 mg/dl
* Fasting blood triglycerides greater than 199 mg/dl
* Fasting blood glucose greater than 109 mg/dl and HbA1c greater than 6.0%
* Individuals currently taking any of the following medications:

  1. blood pressure lowering medication (e.g., beta blockers, ACE inhibitors, angiotensin antagonists, calcium channel blockers, diuretics)
  2. lipid-lowering medication (e.g., statins)
  3. nitrates (e.g. nitroglycerin) for angina
  4. phosphodiesterase inhibitors (e.g., Viagra)
  5. anti-inflammatory drugs
* Individuals currently taking hormone replacement therapy

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N Proctor, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 healthy postmenopausal women were screened for eligibility between October 15, 2013 and January 1, 2020 at State College community in State College, PA.
Pre-assignment Details: 16 of 20 participants were randomized. Of those not randomized, 3 did not meet inclusion criteria and 1 withdrew after the familiarization visit.
Groups:
- Nitrate Depleted Beetroot Juice First, Then Nitrate Rich Beetroot Juice: Subjects consumed 140 ml of beetroot juice (Beet-It Organic Shot) approximately 90 min before physiological testing.
  Nitrate-depleted Beetroot juice (placebo): This beverage is identical in look and taste to the Beet-It organic shot, but has the nitrate removed. It is also bottled and supplied by James White Drinks (UK).
  Nitrate-rich Beetroot juice: This beverage contains 0.3 g of inorganic nitrate per 70 ml container, and is bottled and supplied by James White Drinks (UK).
- Nitrate Rich Beetroot Juice First, Then Nitrate Depleted Beetroot Juice: Subjects consumed 140 ml of beetroot juice (Beet-It Organic Shot) approximately 90 min before physiological testing.
  Nitrate-rich Beetroot juice: This beverage contains 0.3 g of inorganic nitrate per 70 ml container, and is bottled and supplied by James White Drinks (UK).
  Nitrate-depleted Beetroot juice (placebo): This beverage is identical in look and taste to the Beet-It organic shot, but has the nitrate removed. It is also bottled and supplied by James White Drinks (UK).
Period: First Intervention (1day)
Arm/Group | Nitrate Depleted Beetroot Juice First, Then Nitrate Rich Beetroot Juice | Nitrate Rich Beetroot Juice First, Then Nitrate Depleted Beetroot Juice
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout (>7days)
Arm/Group | Nitrate Depleted Beetroot Juice First, Then Nitrate Rich Beetroot Juice | Nitrate Rich Beetroot Juice First, Then Nitrate Depleted Beetroot Juice
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention (1day)
Arm/Group | Nitrate Depleted Beetroot Juice First, Then Nitrate Rich Beetroot Juice | Nitrate Rich Beetroot Juice First, Then Nitrate Depleted Beetroot Juice
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a crossover study.
Groups:
- Randomized, Nitrate-rich or -Depleted Beetroot Juice on Two Separate Days: Subjects consumed 140 ml of beetroot juice (Beet-It Organic Shot) approximately 90 min before physiological testing.
  Nitrate-rich Beetroot juice: This beverage contains 0.3 g of inorganic nitrate per 70 ml container, and is bottled and supplied by James White Drinks (UK).
  Nitrate-depleted Beetroot juice (placebo): This beverage is identical in look and taste to the Beet-It organic shot, but has the nitrate removed. It is also bottled and supplied by James White Drinks (UK).
Arm/Group | Randomized, Nitrate-rich or -Depleted Beetroot Juice on Two Separate Days
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: year] | 63 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Mean arterial pressure [Mean (Full Range); unit: mmHg] | 91 [76 to 110]

OUTCOME MEASURES:

1. Primary Outcome: Resting Aortic Blood Pressures
Description: Aortic Blood pressures were measured in the arm (cuff) and estimated in the aorta (radial artery tonometry).
Time Frame: Resting systolic blood pressure at 90 minutes after beetroot juice ingestion
Population: This was a crossover study where the same group of subjects was intervened with both nitrate-rich beetroot juice and nitrate depleted beetroot juice
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Randomized, Nitrate Rich Beetroot Juice: Subjects consumed 140 ml of beetroot juice (Beet-It Organic Shot) approximately 90 min before physiological testing.
  Beetroot juice: This beverage contains 0.3 g of inorganic nitrate per 70 ml container, and is bottled and supplied by James White Drinks (UK).
- Randomized, Nitrate Depleted Beetroot Juice: Subjects consumed 140 ml of beetroot juice (Beet-It Organic Placebo) approximately 90 min before physiological testing.
  Beetroot juice placebo: This beverage is identical in look and taste to the Beet-It organic shot, but has the nitrate removed. It is also bottled and supplied by James White Drinks (UK).
Arm/Group | Randomized, Nitrate Rich Beetroot Juice | Randomized, Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 13 | 13
mmHg | 113.3 (4.1) | 116.9 (6.3)

2. Secondary Outcome: Blood Measures of Nitrate Absorption and Conversion
Description: Venous blood will be withdrawn (venipuncture) for determination of plasma nitrate and nitrite.
Time Frame: Change from baseline measures of plasma nitrate and nitrite at 90 minutes and at approximately 6 hours
Population: This study is a crossover study. Same subjects for nitrate-rich beetroot juice were intervened for nitrate-depleted beetroot juice.
Measure: Mean (Standard Error); unit: uM
Arm/Group | Randomized, Nitrate Rich Beetroot Juice | Randomized, Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 13 | 13
uM
  Plasma nitrate concentration | 643.9 (45.7) | 39.2 (9.3)
  Plasma Nitrite concentration | 0.402 (0.077) | 0.115 (0.027)

3. Secondary Outcome: Resting Arterial Stiffness/Wave Properties
Description: Carotid to femoral artery pulse wave velocity will be assessed using arterial tonometry.
Time Frame: Change from baseline resting pulse wave velocity at 90 minutes after beet root juice ingestion
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Randomized, Nitrate Rich Beetroot Juice | Randomized, Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 13 | 13
m/s | 7.328 (0.407) | 7.572 (0.384)

4. Secondary Outcome: Handgrip Exercise Blood Pressure Responses (Relative Change From Baseline)
Description: Beat-to-beat blood pressure (finger cuff) will be assessed at rest and during handgrip exercise to volitional fatigue.
Time Frame: Approximately 180 minutes after ingestion of beetroot juice
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Randomized, Nitrate Rich Beetroot Juice | Randomized, Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 8 | 8
percentage of change from baseline | 25 (3) | 30 (5)

5. Secondary Outcome: Peak Rate of Perceived Exertion Scores During Handgrip Exercise
Description: The Borg Rating of Perceived Exertion Scale (RPE) was used to assess exercise intensity during handgrip exercise. The RPE scale ranges from a minimum of 6 (no exertion at all) to a maximum of 20 (maximal exertion) units on a scale.
Time Frame: Approximately 90 minutes after ingestion of beetroot juice
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized, Nitrate Rich Beetroot Juice | Randomized, Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 13 | 13
units on a scale | 17.3 (2.8) | 17.7 (1.7)

6. Secondary Outcome: Handgrip Exercise Tolerance
Description: Time to fatigue (seconds) was assessed during a progressive blood flow restricted handgrip exercise protocol.
Time Frame: Approximately 90 minutes after ingestion of beetroot juice
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Randomized, Nitrate Rich Beetroot Juice | Randomized, Nitrate Depleted Beetroot Juice
Number analyzed (Participants) | 13 | 13
seconds | 602.8 (48.61) | 541.0 (48.66)

ADVERSE EVENTS:
Time Frame: 4 years
Description: not different from the clinicaltrials.gov definitions.
Arm/Group | Randomized, Nitrate Rich Beetroot Juice | Randomized, Nitrate Depleted Beetroot Juice
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT03380000/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT03380000/ICF_001.pdf